CLINICAL TRIAL: NCT04566666
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy And Safety of SCD-044 in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: To Assess the Effect of SCD-044 Treatment on Moderate to Severe Plaque Psoriasis
Acronym: SOLARES-PsO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCD-044-19-14
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo of SCD-044 product (Placebo Comparator): Placebo of SCD-044 study drug
  Interventions: Drug: Placebo
- SCD-044 Tablets_Low Dose (Dose 1) (Active Comparator): SCD-044 tablets at Low Dose (Dose 1)
  Interventions: Drug: SCD-044_Low Dose (Dose 1)
- SCD-044 Tablets_Intermediate Dose (Dose 2) (Active Comparator): SCD-044 tablets at Intermediate Dose (Dose 2)
  Interventions: Drug: SCD-044_Intermediate Dose (Dose 2)
- SCD-044 Tablets_High Dose (Dose 3) (Active Comparator): SCD-044 tablets at High Dose (Dose 3)
  Interventions: Drug: SCD-044_High Dose (Dose 3)

INTERVENTIONS:
Drug: Placebo — Placebo of SCD-044 product
  Arms: Placebo of SCD-044 product
Drug: SCD-044_Low Dose (Dose 1) — SCD-044 tablets in Low Dose (Dose 1)
  Arms: SCD-044 Tablets_Low Dose (Dose 1)
Drug: SCD-044_Intermediate Dose (Dose 2) — SCD-044 tablets in Intermediate Dose (Dose 2)
  Arms: SCD-044 Tablets_Intermediate Dose (Dose 2)
Drug: SCD-044_High Dose (Dose 3) — SCD-044 in High Dose (Dose 3)
  Arms: SCD-044 Tablets_High Dose (Dose 3)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to determine the effect of SCD-044 in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant non-lactating females with a diagnosis of predominantly plaque psoriasis for ≥ 6 months as determined by subject interview and confirmation of diagnosis through physical examination by Investigator.
2. Aged at least 18 years.
3. Subjects with no history of active TB or symptoms of TB

Exclusion Criteria:

1. Subjects with non-plaque forms of psoriasis-like erythrodermic psoriasis, pustular psoriasis, medication-induced, or medication exacerbated psoriasis or new-onset guttate psoriasis.
2. Subjects who have anticipated the requirement of topical therapy, phototherapy, or systemic therapy for psoriasis during the trial.
3. Subjects with history or presence of uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (29):
  - Yuma Clinical Trials, LLC, Yuma, Arizona
  - T. Joseph Raoof Md, Imc./Encino Research Center, Encino, California
  - Metropolis Dermatology, Los Angeles, California
  - Axis Clinical Trials, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Accel Research Sites Network - Annexus Dermatology & Aestheitcs, DeLand, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - Revival Research Corporation, Doral, Florida
  - FXM Clinical Research Fort Lauderdale, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Evolution Clinical Trials, Inc, Hialeah Gardens, Florida
  - JD Medical Group, LLC, Miami, Florida
  - MedOne Clinical Research, LLC, Miami, Florida
  - Century Research LLC, Miami, Florida
  - FXM Clinical Research Miami, Miami, Florida
  - FXM Clinical Research Miramar, Miramar, Florida
  - Adtremed Inc, Tampa, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Oracle Clinical Research, College Park, Georgia
  - Physicians Research Group, West Lafayette, Indiana
  - Revival research Institute, LLC, Troy, Michigan
  - DFW Clinical Research, LLC, Dallas, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Stride Clinical Research, Sugar Land, Texas
  - Springville Dermatology/ CCT Research, Springville, Utah
  - Skin DC Derm, Arlington, Virginia
- El Salvador (3):
  - Clinica de Dermatologia y Cirugia de Piel, La Libertad
  - Clinica Dermatologica, San Salvador
  - Clinica Vargas, San Salvador
- Estonia (2):
  - North Estonia Medical Centre Foundation Ltd., Tallinn
  - Clinical Research Centre OU, Tartu
- Georgia (7):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LLC, Tbilisi
  - Israeli - Georgian Medical Research Clinic Helsikor LLC, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze LLC, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - TIM - Tbilisi Institute of Medicine LLC, Tbilisi
  - David Abuladze Georgian-Italian Clinic LLC, Tbilisi
- Poland (9):
  - ClinicMed, Bialystok
  - Synexus Polska Sp. z o.o. Branch in Gdansk, Gdansk
  - Dobry Lekarz' Modern Therapies Center Limited Liability Company, Krakow
  - Landa Specialist Doctor's Offices, Krakow
  - GLOBE Clinical Research, Kłodzko
  - Appletreeclinics Clinical Research Centre, Lodz
  - EMC Medical Institute Joint Stock Company, "Certus" Private Healthcare Facility Hospital No. 1, Poznan
  - TWOJA PRZYCHODNIA Medical Centre of Szczecin, Twoja Przychodnia SCM, Szczecin
  - National Medical Institute of the MSWiA, Clinical Department of Dermatology, Warsaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Participant Flow is based on the safety population
Groups:
- Part 1- Placebo of SCD-044 Product: Placebo of SCD-044 study drug
  Placebo: Placebo of SCD-044 product
- Part 1- SCD-044 Tablets_Low Dose (Dose 1): SCD-044 tablets at Low Dose (Dose 1)
  SCD-044_Dose 1: SCD-044 tablets in Low Dose (Dose 1)
- Part 1- SCD-044 Tablets_Intermediate Dose (Dose 2): SCD-044 tablets at Intermediate Dose (Dose 2)
  SCD-044_Dose 2: SCD-044 tablets in Intermediate Dose (Dose 2)
- Part 1- SCD-044 Tablets_High Dose (Dose 3): SCD-044 tablets at High Dose (Dose 3)
  SCD-044_Dose 3: SCD-044 in High Dose (Dose 3)
- Part 2- Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Part I (16 weeks)- Placebo; Part II (Week 16 to Week 28:)- Part I responders will be re-randomized to SCD-044 tablets of intermediate dose (Dose 2)
- Part 2- Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3): Part 1- Placebo Part 2- Part I responders will be re-randomized to SCD-044 tablets of high dose (Dose 3)
- Part 2- Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1): Part 1- SCD-044 tablets of low dose (Dose 2) Part 2- Part I responders will remain on SCD-044 tablets of low dose (Dose 1)
- Part 2- Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2): Part 1- SCD-044 tablets of intermediate dose (Dose 2) Part 2- Part I responders will remain on SCD-044 tablets of intermediate dose (Dose 2)
- Part 2- Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3): Part 1- SCD-044 tablets of high dose (Dose 3) Part 2- Part I responders will remain on SCD-044 tablets of high dose (Dose 3)
- Part 2- Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2): Part 1- Placebo Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of intermediate dose (Dose 2)
- Part 2- Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3): Part 1- Placebo Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3)
- Part 2- Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3): Part 1- SCD-044 tablets of low dose (Dose 2) Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3)
- Part 2- Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3): Part 1- SCD-044 tablets of intermediate dose (Dose 2) Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3)
Period: Part 1
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1- SCD-044 Tablets_Low Dose (Dose 1) | Part 1- SCD-044 Tablets_Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets_High Dose (Dose 3) | Part 2- Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part 2- Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part 2- Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part 2- Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part 2- Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part 2- Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part 2- Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Started | 64 | 71 | 69 | 59 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 49 | 59 | 57 | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 12 | 12 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1- SCD-044 Tablets_Low Dose (Dose 1) | Part 1- SCD-044 Tablets_Intermediate Dose (Dose 2) | Part 1- SCD-044 Tablets_High Dose (Dose 3) | Part 2- Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part 2- Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part 2- Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part 2- Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part 2- Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part 2- Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part 2- Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part 2- Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part 2- Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Started | 0 | 0 | 0 | 0 | 9 | 12 | 32 | 36 | 45 | 10 | 15 | 25 | 21
Completed | 0 | 0 | 0 | 0 | 8 | 11 | 30 | 33 | 20 | 7 | 8 | 20 | 15
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 25 | 3 | 7 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- SCD-044 Tablets_Dose 1: SCD-044_Dose 1: SCD-044 tablets in Dose 1.
- SCD-044 Tablets_Dose 2: SCD-044_Dose 2: SCD-044 tablets in Dose 2
- SCD-044 Tablets_Dose 3: SCD-044_Dose 3: SCD-044 in Dose 3
- Total: Total of all reporting groups
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3 | Total
Number analyzed (Participants) | 64 | 71 | 69 | 59 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.99) | 44.8 (13.87) | 46.3 (13.63) | 46.3 (13.43) | 46.2 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 24 | 27 | 100
  Male | 42 | 44 | 45 | 32 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6 | 12
  White | 61 | 60 | 61 | 52 | 234
  More than one race | 0 | 8 | 6 | 1 | 15
  Other | 0 | 1 | 0 | 0 | 1
  Hispanic or Latino | 43 | 31 | 31 | 42 | 147
  Not Hispanic or Latino | 21 | 40 | 38 | 17 | 116

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With at Least 75% Improvement in PASI (PASI 75)
Description: The subjects showing at least 75% improvement in Psoriasis Area and Severity Index score on a scale of 0-4 score. Higher score denotes more severe disease activity.
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week16
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 50 | 60 | 61 | 48
percentage of subjects | 14.0 | 28.3 | 23.0 | 16.7
Statistical Analysis 1: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 1; Test type: Superiority; p = 0.1011, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 2; Test type: Superiority; p = 0.2666, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 3; Test type: Superiority; p = 0.7394, Cochran-Mantel-Haenszel

2. Secondary Outcome: Investigator's Global Assessment (IGA) Score
Description: The subjects achieving predefined improvement (0 or 1) in Investigator's Global Assessment (IGA) of disease severity on a scale of 0 to 4 score with at least two-grade reduction from Baseline to Week 16. 0 indicates clear, while 1 indicates almost clear, while 4 is severe.
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week 16
Measure: Number; unit: percentage of subject
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 50 | 60 | 61 | 48
percentage of subject | 0 | 10.0 | 9.8 | 8.3
Statistical Analysis 1: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 1; Test type: Superiority; p = 0.1376, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 2; Test type: Superiority; p = 0.1254, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo of SCD-044 Product vs SCD-044 Tablets_Dose 3; Test type: Superiority; p = 0.2349, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: The subjects achieving predefined improvement in Psoriasis Area and Severity Index (PASI) on a scale of 0-4 score. Higher score denotes more severe disease activity..
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2): Part I (16 weeks)- Placebo Part II (Week 16 to Week 28:)- Part I responders will be re-randomized to SCD-044 tablets of intermediate dose (Dose 2) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3): Part 1- Placebo Part 2- Part I responders will be re-randomized to SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1): Part 1- SCD-044 tablets of low dose (Dose 2) Part 2- Part I responders will remain on SCD-044 tablets of low dose (Dose 1) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2): Part 1- SCD-044 tablets of intermediate dose (Dose 2) Part 2- Part I responders will remain on SCD-044 tablets of intermediate dose (Dose 2) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3): Part 1- SCD-044 tablets of high dose (Dose 3) Part 2- Part I responders will remain on SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2): Part 1- Placebo Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of intermediate dose (Dose 2) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3): Part 1- Placebo Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3): Part 1- SCD-044 tablets of low dose (Dose 2) Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
- Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3): Part 1- SCD-044 tablets of intermediate dose (Dose 2) Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 26 | 27 | 20 | 2 | 3 | 9 | 6
score on a scale | -3.58 (1.813) | -2.03 (5.069) | -17.18 (7.685) | -16.12 (4.338) | -17.11 (6.570) | -9.30 (2.970) | -20.87 (16.686) | -10.58 (5.401) | -11.62 (6.010)

4. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Response Rate
Description: Psoriasis Area and Severity Index (PASI50, PASI75, PASI90, and PASI100) response rate at Week 16.
  PASI50, PASI75, PASI90 and PASI100 are defined as 50%, 75%, 90% and 100% decrease from baseline in PASI correspondingly.
  The data represents the percentage of subject who achieved PASI 50, PASI 75, PASI 90, and PASI 100 at week 16.
Time Frame: Week 16
Measure: Number; unit: Percentage of subject
Groups:
- Placebo of SCD-044 Product: Placebo tablet of SCD-044 product
- SCD-044 Tablets_Dose 1: SCD-044 Tablets of low dose (Dose 1)
- SCD-044 Tablets_Dose 2: SCD-044 Tablets of intermediate dose (Dose 2)
- SCD-044 Tablets_Dose 3: SCD-044 Tablets of high dose (Dose 3)
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 49 | 59 | 57 | 46
Percentage of subject
  PASI 50 | 46.9 | 47.5 | 56.1 | 50.0
  PASI 75 | 14.3 | 28.8 | 26.3 | 17.4
  PASI 90 | 0 | 6.8 | 7.0 | 2.2
  PASI 100 | 0 | 3.4 | 1.8 | 2.2
Statistical Analysis 1: Comparison: Placebo of SCD-044 Product; The data represents the Statistical Analysis for PASI 100; Test type: Superiority; Binomial proportion = 0, 95% CI 2-sided [0.0 to 7.3]
Statistical Analysis 2: Comparison: SCD-044 Tablets_Dose 1; The data represents the Statistical Analysis for PASI 100; Test type: Superiority; binomial proportion = 3.4, 95% CI 2-sided [0.4 to 11.7]
Statistical Analysis 3: Comparison: SCD-044 Tablets_Dose 2; The data represents the Statistical Analysis for PASI 100; Test type: Superiority; binomial proportion = 1.8, 1.8% CI 2-sided [0.0 to 9.4]
Statistical Analysis 4: Comparison: SCD-044 Tablets_Dose 3; The data represents the Statistical Analysis for PASI 100; Test type: Superiority; binomial proportion = 2.2, 95% CI 2-sided [0.1 to 11.5]
Statistical Analysis 5: Comparison: Placebo of SCD-044 Product; The data represents the Statistical Analysis for PASI 50; Test type: Superiority; binomial proportion = 46.9, 95% CI 2-sided [32.5 to 61.7]
Statistical Analysis 6: Comparison: SCD-044 Tablets_Dose 1; The data represents the Statistical Analysis for PASI 50; Test type: Superiority; binomial proportion = 47.5, 95% CI 2-sided [34.3 to 60.9]
Statistical Analysis 7: Comparison: SCD-044 Tablets_Dose 2; The data represents the Statistical Analysis for PASI 50; Test type: Superiority; binomial proportion = 56.1, 95% CI 2-sided [42.4 to 69.3]
Statistical Analysis 8: Comparison: SCD-044 Tablets_Dose 3; The data represents the Statistical Analysis for PASI 50; Test type: Superiority; binomial proportion = 50.0, 95% CI 2-sided [34.9 to 65.1]
Statistical Analysis 9: Comparison: Placebo of SCD-044 Product; The data represents the Statistical Analysis for PASI 75; Test type: Superiority; binomial proportion = 14.3, 95% CI 2-sided [5.9 to 27.2]
Statistical Analysis 10: Comparison: SCD-044 Tablets_Dose 1; The data represents the Statistical Analysis for PASI 75; Test type: Superiority; binomial proportion = 28.8, 95% CI 2-sided [17.8 to 42.1]
Statistical Analysis 11: Comparison: SCD-044 Tablets_Dose 2; The data represents the Statistical Analysis for PASI 75; Test type: Superiority; binomial proportion = 26.3, 95% CI 2-sided [15.5 to 39.7]
Statistical Analysis 12: Comparison: SCD-044 Tablets_Dose 3; The data represents the Statistical Analysis for PASI 75; Test type: Superiority; binomial proportion = 17.4, 95% CI 2-sided [7.8 to 31.4]
Statistical Analysis 13: Comparison: Placebo of SCD-044 Product; The data represents the Statistical Analysis for PASI 90; Test type: Superiority; binomial proportion = 0.0, 95% CI 2-sided [0.0 to 7.3]
Statistical Analysis 14: Comparison: SCD-044 Tablets_Dose 1; The data represents the Statistical Analysis for PASI 90; Test type: Superiority; binomial proportion = 6.8, 95% CI 2-sided [1.9 to 16.5]
Statistical Analysis 15: Comparison: SCD-044 Tablets_Dose 2; The data represents the Statistical Analysis for PASI 90; Test type: Superiority; binomial proportion = 7.0, 95% CI 2-sided [1.9 to 17.0]
Statistical Analysis 16: Comparison: SCD-044 Tablets_Dose 3; The data represents the Statistical Analysis for PASI 90; Test type: Superiority; binomial proportion = 2.2, 95% CI 2-sided [0.1 to 11.5]

5. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Response Rate
Description: Psoriasis Area and Severity Index (PASI50, PASI75, PASI90, and PASI100) response rate at Week 52 The data represents the percentage of subject who achieved PASI 50, PASI 75, PASI 90, and PASI 100 at week 16.
Time Frame: Week 52
Measure: Number; unit: percentage of subjects
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 26 | 27 | 20 | 2 | 3 | 9 | 6
percentage of subjects
  PASI 50 | 66.7 | 66.7 | 88.5 | 92.6 | 95.0 | 50.0 | 100.0 | 88.9 | 100.0
  PASI 75 | 33.3 | 44.4 | 84.6 | 66.7 | 90.0 | 0 | 66.7 | 66.7 | 83.3
  PASI 90 | 16.7 | 11.1 | 46.2 | 33.3 | 55.0 | 0 | 0 | 0 | 16.7
  PASI 100 | 0 | 0 | 7.7 | 3.7 | 10.0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Psoriasis Symptoms and Signs Diary (PSSD) at Week 16
Description: At study week 0, 16, and 52; based on 11-item questionnaire, the symptoms and patient-observable signs in psoriasis will be scored using 0 to 10 rating scale (0-absent, 10-worst imaginable). The summary score is the sum of item scores (0-110), and a higher score indicates more severe disease- 0- best outcome 110- worst outcome
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 49 | 59 | 57 | 46
score on a scale | -19.5 (28.75) | -23.2 (28.42) | -23.8 (26.58) | -23.6 (28.69)

7. Secondary Outcome: Change From Baseline in Psoriasis Symptoms and Signs Diary (PSSD) at Week 52
Description: as for outcome 6
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 25 | 27 | 20 | 2 | 3 | 9 | 6
score on a scale | -7.0 (10.08) | -9.6 (17.21) | -35.0 (18.94) | -33.6 (25.03) | -55.7 (20.87) | -26.0 (59.40) | -24.0 (23.07) | -12.7 (34.29) | -20.8 (19.75)

8. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: At study week 0, 16, and 52; based on 10-item questionnaire on skin problems (0 to 3 scale).
  The scoring of each question is as follows: Very Much or Yes = 3, A lot = 2, A little = 2, Not relevant or Not at all or No = 0.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  Total score range: 0-30 (higher = greater impact).
  Interpretation bands:
  0-1: No effect 2-5: Small effect 6-10: Moderate effect 11-20: Very large effect 21-30: Extremely large effect.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 49 | 59 | 57 | 46
score on a scale | -5.0 (7.00) | -4.0 (6.58) | -4.6 (6.50) | -4.4 (6.50)

9. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 52
Description: as for outcome 8
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 25 | 27 | 20 | 2 | 3 | 9 | 6
score on a scale | -1.5 (1.22) | -2.9 (3.72) | -7.8 (5.28) | -6.2 (5.88) | -10.7 (4.00) | -2.5 (4.95) | -3.0 (6.24) | -4.6 (6.27) | -4.2 (4.54)

10. Secondary Outcome: Investigator's Global Assessment (IGA) Score
Description: The subjects achieving predefined improvement (0 or 1) in Investigator's Global Assessment (IGA) of disease severity on a scale of 0 to 4 score with at least two-grade reduction from Baseline to Week 52. 0 indicates clear, while 1 indicates almost clear, while 4 is severe.
  The information presented represents the percentage of subjects, calculated as the proportion of subjects multiplied by 100.
Time Frame: Week 52
Measure: Number; unit: Percentage of participants
Groups:
- Part I Non-Responders:SCD-044 Low Dose (Dose 1) to High Dose (Dose 3): Part 1- SCD-044 tablets of low dose (Dose 2) Part 2- Part I non-responders will be re-randomized to SCD-044 tablets of high dose (Dose 3) Part III (Week 28 to Week 52): Part II non-responder will be discontinued from the study and responders will continue their existing dosing regimen until the end of Part III.
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders:SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 26 | 27 | 20 | 2 | 3 | 9 | 6
Percentage of participants | 16.7 | 11.1 | 38.5 | 44.4 | 65.0 | 0 | 0 | 22.2 | 0

11. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) at Week 16
Description: At study weeks 16, and 52, the Investigator will assess % BSA affected with psoriasis.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 49 | 59 | 57 | 46
% BSA | -7.21 (9.608) | -8.32 (16.194) | -9.57 (12.983) | -9.63 (12.794)

12. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) at Week 52
Description: At study weeks 16, and 52, the Investigator will assess % BSA affected with psoriasis.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 26 | 27 | 20 | 2 | 3 | 9 | 6
% BSA | -7.17 (5.913) | -11.01 (9.658) | -21.60 (12.206) | -21.77 (13.283) | -26.03 (13.368) | -12.50 (2.121) | -25.67 (26.652) | -19.00 (13.285) | -15.17 (16.666)

13. Secondary Outcome: Patient Global Impression of Severity (PGIS)
Description: Subjects will be asked to assess their overall impression of disease severity using a scale of None, Mild, Moderate or Severe (None- best outcome no symptoms; Severe- worst symptoms)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 63 | 71 | 68 | 59
Participants
  None | 0 | 0 | 0 | 1
  Mild | 4 | 4 | 2 | 1
  Moderate | 31 | 35 | 44 | 36
  Severe | 28 | 32 | 22 | 21

14. Secondary Outcome: Patient Global Impression of Severity (PGIS)
Description: At study weeks 0, 16, and 52, subjects will be asked to assess their overall impression of disease severity using a scale of None, Mild, Moderate or Severe.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo of SCD-044 Product | SCD-044 Tablets_Dose 1 | SCD-044 Tablets_Dose 2 | SCD-044 Tablets_Dose 3
Number analyzed (Participants) | 49 | 59 | 57 | 46
Participants
  None | 1 | 4 | 4 | 3
  Mild | 18 | 20 | 26 | 14
  Moderate | 19 | 29 | 21 | 25
  Severe | 11 | 6 | 6 | 4

15. Secondary Outcome: Patient Global Impression of Severity (PGIS)
Description: Subjects will be asked to assess their overall impression of disease severity using a scale of None, Mild, Moderate or Severe.
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 25 | 27 | 20 | 2 | 3 | 9 | 6
Participants
  None | 0 | 2 | 3 | 2 | 6 | 0 | 0 | 0 | 0
  Mild | 6 | 4 | 15 | 15 | 12 | 1 | 3 | 6 | 5
  Moderate | 0 | 3 | 6 | 9 | 2 | 1 | 0 | 3 | 1
  Severe | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Subjects will be asked to assess if there has been a change in clinical status using a 5 point scale (1 to 5). 1 indicating 'Much better', while 5 indicating 'Much Worse'.
Time Frame: Week 52
Measure: Number; unit: participants
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders: SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 9 | 25 | 27 | 20 | 2 | 3 | 9 | 6
participants
  Much Better | 5 | 6 | 15 | 13 | 18 | 1 | 2 | 2 | 2
  A Little Better | 1 | 3 | 5 | 9 | 2 | 1 | 1 | 5 | 3
  No Change | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 2 | 1
  A Little Worse | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Much Worse | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Evaluate Pharmacokinetic Parameter
Description: Steady-state maximum plasma concentration (Cmax-ss)
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part I Responders: Placebo to SCD-044 Tablets of Intermediate Dose (Dose 2) | Part I Responders: Placebo to SCD-044 Tablets of High Dose (Dose 3) | Part I Responders: SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | Part I Responders: SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | Part I Responders: SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | Part I Non-Responders: Placebo to SCD-044 Intermediate Dose (Dose 2) | Part I Non-Responders: Placebo to SCD-044 High Dose (Dose 3) | Part I Non-Responders:SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | Part I Non-Responders: SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 6 | 8 | 24 | 27 | 18 | 2 | 3 | 9 | 6
pg/mL | 3242.187 (3944.1894) | 1928.714 (3388.7518) | 2528.022 (2934.3946) | 3065.187 (2612.9302) | 3309.121 (4368.2414) | 2831.310 (4004.0770) | 5941.477 (6859.1232) | 7264.772 (6296.6163) | 4197.117 (4724.9842)

18. Secondary Outcome: Subjects With Adverse Events
Description: Total Number Affected by adverse events from Baseline through Week 56
Time Frame: Week 56
Measure: Count of Participants; unit: Participants
Groups:
- Part 1- Placebo of SCD-044 Product: Placebo tablet of SCD-044 product
- Part 1- SCD-044 Tablets_Dose 1: SCD-044 Tablets of low dose (Dose 1)
- Part 1- SCD-044 Tablets_Dose 2: SCD-044 Tablets of intermediate dose (Dose 2)
- Part 1- SCD-044 Tablets_Dose 3: SCD-044 Tablets of high dose (Dose 3)
- Placebo to SCD-044 Intermediate Dose (Dose 2): Subjects initially randomized to Placebo re-randomized to SCD-044 tablets of intermediate dose in Part II
- Placebo to SCD-044 High Dose (Dose 3): Subjects initially randomized to Placebo re-randomized to SCD-044 tablets of high dose in Part II
- SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1): Subjects initially randomized to SCD-044 low dose continue the same treatment in part II
- SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2): Subjects initially randomized to SCD-044 intermediate dose continue the same treatment in part II
- SCD-044 High Dose (Dose 3) to High Dose (Dose 3): Subjects initially randomized to SCD-044 high dose continue the same treatment in part II
- SCD-044 Low Dose (Dose 1) to High Dose (Dose 3): Subjects initially randomized to low dose re-randomized to SCD-044 tablets of high dose in Part II
- SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3): Subjects initially randomized to intermediate dose re-randomized to SCD-044 tablets of high dose in Part II
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1- SCD-044 Tablets_Dose 1 | Part 1- SCD-044 Tablets_Dose 2 | Part 1- SCD-044 Tablets_Dose 3 | Placebo to SCD-044 Intermediate Dose (Dose 2) | Placebo to SCD-044 High Dose (Dose 3) | SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
Number analyzed (Participants) | 64 | 71 | 69 | 59 | 18 | 22 | 32 | 36 | 20 | 20 | 16
Participants
  Subjects with serious TEAE | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects with any TEAE | 17 | 26 | 27 | 18 | 4 | 3 | 14 | 13 | 9 | 6 | 1

ADVERSE EVENTS:
Time Frame: 56 Weeks
Arm/Group | Part 1- Placebo of SCD-044 Product | Part 1- SCD-044 Tablets_Dose 1 | Part 1- SCD-044 Tablets_Dose 2 | Part 1- SCD-044 Tablets_Dose 3 | Placebo to SCD-044 Intermediate Dose (Dose 2) | Placebo to SCD-044 High Dose (Dose 3) | SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) | SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) | SCD-044 High Dose (Dose 3) to High Dose (Dose 3) | SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) | SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/71 | 0/69 | 0/59 | 0/18 | 0/22 | 0/32 | 0/36 | 0/20 | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/71 | 2/69 | 0/59 | 0/18 | 0/22 | 0/32 | 0/36 | 0/20 | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 17/64 | 26/71 | 27/69 | 18/59 | 4/18 | 3/22 | 14/32 | 13/36 | 9/20 | 6/20 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Placebo of SCD-044 Product (N=64) | Part 1- SCD-044 Tablets_Dose 1 (N=71) | Part 1- SCD-044 Tablets_Dose 2 (N=69) | Part 1- SCD-044 Tablets_Dose 3 (N=59) | Placebo to SCD-044 Intermediate Dose (Dose 2) (N=18) | Placebo to SCD-044 High Dose (Dose 3) (N=22) | SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) (N=32) | SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) (N=36) | SCD-044 High Dose (Dose 3) to High Dose (Dose 3) (N=20) | SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) (N=20) | SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3) (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part 1- Placebo of SCD-044 Product (N=64) | Part 1- SCD-044 Tablets_Dose 1 (N=71) | Part 1- SCD-044 Tablets_Dose 2 (N=69) | Part 1- SCD-044 Tablets_Dose 3 (N=59) | Placebo to SCD-044 Intermediate Dose (Dose 2) (N=18) | Placebo to SCD-044 High Dose (Dose 3) (N=22) | SCD-044 Low Dose (Dose 1) to Low Dose (Dose 1) (N=32) | SCD-044 Intermediate Dose (Dose 2) to Intermediate Dose (Dose 2) (N=36) | SCD-044 High Dose (Dose 3) to High Dose (Dose 3) (N=20) | SCD-044 Low Dose (Dose 1) to High Dose (Dose 3) (N=20) | SCD-044 Intermediate Dose (Dose 2) to High Dose (Dose 3) (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinoatrial block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 2 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Penile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 5 | 2 | 2 | 0 | 0 | 1 | 3 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 4 | 2 | 3 | 0 | 0 | 2 | 0 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0/0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04566666/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04566666/SAP_001.pdf